CLINICAL TRIAL: NCT03767842
Title: Volumetric Impedance to Guide Stroke Response
Acronym: VIGOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cerebrotech Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CH007
Record Dates: First submitted 2018-12-03; First posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Visor System — Subjects are monitored one time with the Visor System.

SUMMARY:
Assess the ability of the Visor System to detect hemispheric bioimpedance asymmetry

ELIGIBILITY:
Inclusion Criteria:

* Being evaluated as a suspected stroke

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients presenting for evaluation of acute stroke
Sampling Method: Non-Probability Sample
Enrollment: 316 (Estimated)
Dates: Start 2018-07-18 (Actual); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Hemispheric bioimpedance asymmetry sensitivity and specificity | At the time of device monitoring - day 0
  Ability of the device to detect bioimpedance asymmetry in patients presenting with symptoms of acute stroke

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Kellner, MD, Principal Investigator — Sinai Health System; Andrei V Alexandrov, MD, Principal Investigator — University of Tennessee; Raul G Nogueira, MD, Principal Investigator — Emory University School of Medicine, Grady Memorial Hospital
Locations (1):
- University of Buffalo Neurosurgery, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kellner CP, Sauvageau E, Snyder KV, Fargen KM, Arthur AS, Turner RD, Alexandrov AV. The VITAL study and overall pooled analysis with the VIPS non-invasive stroke detection device. J Neurointerv Surg. 2018 Nov;10(11):1079-1084. doi: 10.1136/neurintsurg-2017-013690. Epub 2018 Mar 6. PMID 29511114